CLINICAL TRIAL: NCT07136636
Title: Investigating the Prognostic Accuracy of Different Biomarkers for Detection of Developmental Language Disorder in Children With Neonatal Encephalopathy
Brief Title: Speech of Kids After Neonatal Encephalopathy
Acronym: SANE
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: UiT The Arctic University of Norway (Other); Budapest University of Technology and Economics (Other); Eotvos Lorand University (Other)
Responsible Party: Sponsor
Other Study IDs: NNGYK/24844-9/2025
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIE - Hypoxic - Ischemic Encephalopathy; Language Delay; Autism; ADHD - Attention Deficit Disorder With Hyperactivity; Specific Language Impairment; Intellectual Developmental Disorder
Keywords: HIE - Hypoxic - Ischemic Encephalopathy; delayed language development; neurodevelopment; MRI; biomarker; corpus callosum diffusion restriction; IQ; newborn prediction tool
MeSH Terms: conditions — Language Development Disorders; Autistic Disorder; Attention Deficit Disorder with Hyperactivity; Specific Language Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children born with Hypoxic-Ischemic Encephalopathy (HIE)

SUMMARY:
The goal of this ambispective cohort study is to reveal the early indicators of delayed language development in children born with hypoxic-ischemic encephalopathy (HIE).

We will examine the prognostic accuracy of different biomarkers, with a special focus on the ADC values of the corpus callosum.

The main questions it aims to answer are:

1. To what extent does hypoxic-ischemic encephalopathy (HIE) in infancy affect intellectual development (IQ), receptive and expressive language abilities at different levels of the language system, and memory capacities related to language development?
2. What is the relationship between early biomarkers of brain injury-such as blood gas levels, lactate, aEEG, and MRI findings (Weeke scoring system, ADC values of the corpus callosum)-and long-term cognitive developmental outcomes?
3. What is the incidence of autism spectrum disorder (ASD) and attention deficit hyperactivity disorder (ADHD) in this high-risk population of infants with HIE?
4. Is there an association between the Weeke Total Score and long-term language developmental outcomes?
5. Can restricted diffusion (ADC values) of the splenium of the corpus callosum serve as an early neuroradiological marker of developmental language disorder (DLD)?

Our participants are children born between 2017 and 2023 with moderate to severe HIE, treated with therapeutic hypothermia at Semmelwies University Children's Hospital. During their first days of life, several neonatal measurements were taken (blood gas markers, aEEG etc.), and at day 4-5, they had an MRI scan of their brain. The MRI scans will be reanalyzed, using the Weeke MRI scoring system. These children underwent a neurodevelopmental follow-up at the age of 2 years and currently, they will have another follow-up at the age of 4-7 years.

DETAILED DESCRIPTION:
This ambispective, single-center cohort study will investigate the cognitive and language development of children aged 4-7 years who were previously treated for hypoxic-ischemic encephalopathy (HIE) and underwent standardized neurodevelopmental assessment at two years of age. In addition to developmental outcomes, the study will incorporate clinical, laboratory, and imaging data collected during the neonatal period. All available neonatal MRI scans will be re-evaluated according to predefined criteria. Recruitment and data collection will take place from April 1, 2025, to December 31, 2026. The study population will include children whose parents provided consent for follow-up assessments at the two-year evaluation.

Phase 1.: Blood gas values like pH, base deficit, PCO2, PO2, HCO3, and lactate were registered. aEEG cerebral activity was recorded using continuous single channel (biparietal, P3-P4) aEEG monitoring. It started before 6 hours of age.

Phase 2. : MRI scans was perfomed between the 4-5th day of postnatal age. The MRI scans will be reanalyzed, using the Weeke MRI scoring system.

Phase 3. : At the age of 2 years participating children underwent neurodevelopemntal follow-up, where the Bayley Scales of Infant and Toddler Development, Second Edition (Bayley-II) was used. It is a standardized tool for assessing the developmental functioning of children from 1 to 42 months of age. The test provides both a Mental Development Index (MDI) and a Psychomotor Development Index (PDI) to summarize performance in key areas.

Phase 4.: At the age of 4-7 years the children will undergo their second neurodevelopmental assessment. Within this assessment we will administer the following:

Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI-IV), which assesses Full-Scale IQ, Verbal IQ, and Performance IQ in children aged 4 years to 7 years.

Complex Test of Spoken Language Skills (KOBAK), the first comprehensive, standardized language assessment developed for Hungarian-speaking children. The KOBAK comprises 16 subtests evaluating expressive and receptive language functions across multiple domains (phonology, lexical semantics, morphology, syntax, and pragmatics), as well as speech motor functions and verbal working memory. The test enables evidence-based differentiation of average, above-average, and below-average language abilities; provides a detailed language profile; supports the assessment of school readiness; and facilitates screening, diagnosis, differential diagnosis, and longitudinal monitoring of language development.

As part of the neurodevelopmental assessment, parents will complete several questionnaires:

Socioeconomic Questionnaire (assessing parental education, income, and related variables) Jaworsky Questionnaire Social Communication Questionnaire (SCQ) ScreenQ ADHD Rating Scale Strengths and Difficulties Questionnaire (SDQ)

ELIGIBILITY:
Children born between 2017 and 2023 with moderate to severe HIE, treated with therapeutic hypothermia at Semmelweis University Children's Hospital.

Inclusion criteria

1. Born at ≥ 35th week of gestation
2. Attended follow-up examinations at two years of age
3. Has parental informed consent

Exclusion criteria

1. Hearing loss
2. Multilingual language environment
3. Congenital abnormalities
4. Metabolic disease
5. Sudden unexpected postnatal collapse
6. Brain injury not caused by HIE
7. Severe motor impairment defined as a score <70 on the psychomotor development index (PDI) at 2 years of age

Ages: 0 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with HIE
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive abilities - WPPSI-IV | At the age of 4-7 years
Language abilities - KOBAK | At the age of 4-7 years

SECONDARY OUTCOMES:
Socioeconomic status - Socioeconomic questionnaire | At the age of 4-7 years
Parental concerns - Jaworsky Questionnaire | At the age of 4-7 years
Social and Communication skills - Social Communication Questionnaire | At the age of 4-7 years
Digital screen use - ScreenQ | At the age of 4-7 years
ADHD traits - ADHD Rating Scale | At the age of 4-7 years
Behavior - Strengths and Difficulties Questionnaire | At the age of 4-7 years

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

REFERENCES:
- [Background] Bartha-Doering L, Kollndorfer K, Schwartz E, Fischmeister FPS, Alexopoulos J, Langs G, Prayer D, Kasprian G, Seidl R. The role of the corpus callosum in language network connectivity in children. Dev Sci. 2021 Mar;24(2):e13031. doi: 10.1111/desc.13031. Epub 2020 Sep 1. PMID 32790079
- [Background] Weeke LC, Groenendaal F, Mudigonda K, Blennow M, Lequin MH, Meiners LC, van Haastert IC, Benders MJ, Hallberg B, de Vries LS. A Novel Magnetic Resonance Imaging Score Predicts Neurodevelopmental Outcome After Perinatal Asphyxia and Therapeutic Hypothermia. J Pediatr. 2018 Jan;192:33-40.e2. doi: 10.1016/j.jpeds.2017.09.043. PMID 29246356
- [Background] Ni Bhroin M, Kelly L, Sweetman D, Aslam S, O'Dea MI, Hurley T, Slevin M, Murphy J, Byrne AT, Colleran G, Molloy EJ, Bokde ALW. Relationship Between MRI Scoring Systems and Neurodevelopmental Outcome at Two Years in Infants With Neonatal Encephalopathy. Pediatr Neurol. 2022 Jan;126:35-42. doi: 10.1016/j.pediatrneurol.2021.10.005. Epub 2021 Oct 13. PMID 34736061
- [Background] Chin EM, Jayakumar S, Ramos E, Gerner G, Soares BP, Cristofalo E, Leppert M, Allen M, Parkinson C, Johnston M, Northington F, Burton VJ. Preschool Language Outcomes following Perinatal Hypoxic-Ischemic Encephalopathy in the Age of Therapeutic Hypothermia. Dev Neurosci. 2019 Jun 5:1-11. doi: 10.1159/000499562. Online ahead of print. PMID 31167188
- [Background] Ouwehand S, Smidt LCA, Dudink J, Benders MJNL, de Vries LS, Groenendaal F, van der Aa NE. Predictors of Outcomes in Hypoxic-Ischemic Encephalopathy following Hypothermia: A Meta-Analysis. Neonatology. 2020;117(4):411-427. doi: 10.1159/000505519. Epub 2020 Apr 1. PMID 32235122